CLINICAL TRIAL: NCT00073307
Title: A Phase III Randomized Study of BAY43-9006 in Patients With Unresectable and/or Metastatic Renal Cell Cancer.
Brief Title: Study of BAY43-9006 in Patients With Unresectable and/or Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11213
Record Dates: First submitted 2003-11-19; First posted 2003-11-21 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Cancer (RCC); Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily). Dose modification due to toxicity was permitted.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo (Placebo Comparator): Placebo tablets matching in appearance were to be orally administered twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Multi Kinase Inhibitor
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, efficacy (including quality of life), and pharmacokinetics of BAY43-9006 when added to Best Supportive Care in patients with unresectable and/or metastatic renal cell cancer, who have received one prior systemic regimen for advanced disease.

DETAILED DESCRIPTION:
Overall Survival (OS), Patient-reported outcome (PRO)

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable and/or metastatic, measurable renal cell carcinoma histologically or cytologically documented
* Patients must have had one prior systemic therapy for advanced disease, which was completed at least 30 days but no longer than 8 months prior to randomization
* Patients who have at least one uni-dimensional measurable lesion by CT-scan or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients who have an Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1
* Patients who have adequate coagulation, liver and kidney functions

Exclusion Criteria:

* Patients with rare subtypes of renal cell carcinoma (RCC) such as pure papillary cell tumors, mixed tumor containing predominantly sarcomatoid cells, Bellini carcinoma, medullary carcinoma, or chromophobe oncocytic tumors
* Previous malignancy (except for cervical carcinoma in situ, adequately treated basal cell carcinoma,or superficial bladder tumors, or other malignancies curatively treated > 2 years prior to entry
* Cardiac arrhythmias requiring anti-arrhythmics, symptomatic coronary artery disease or ischemia or congestive heart failure
* Patients with a history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Patients with a history or presence of metastatic brain or meningeal tumors
* Patients with seizure disorder requiring medication (such as anti-epileptics)
* History of organ allograft or bone marrow transplant of stem cell rescue
* Patients who are pregnant or breast-feeding Women of childbearing potential must have a negative pregnancy test prior to drug administration. Both men and women enrolled in this trial must use adequate birth control
* Patients who have three or more of the following:

  * ECOG performance status greater than or equal to 2,
  * Abnormally high lactate dehydrogenase,
  * Abnormally high serum hemoglobin,
  * Abnormally high corrected serum calcium,
  * Absence of prior nephrectomy
* Excluded therapies and medications, previous and concomitant:

  * Concurrent anti-cancer chemotherapy, immunotherapy or hormonal therapy except biphosphonates
  * Significant surgery with 4 weeks of start of study
  * Investigational drug therapy during or within 30 days
  * Concomitant treatment with rifampin or St. John's Wort
  * Prior use of Raf-kinase inhibitors (RKI), MEK or Farnesyl transferase inhibitors
  * Prior use of Bevacizumab, and all other drugs (investigational or licensed) that target VEGF/VEGF receptors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2003-11; Primary Completion 2006-09 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (115):
- United States (30):
  - Tucson, Arizona
  - Los Angeles, California
  - Sacramento, California
  - Aurora, Colorado
  - Hamden, Connecticut
  - Atlanta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Lafayette, Louisiana
  - Frederick, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Brooklyn, New York
  - New York, New York
  - The Bronx, New York
  - Canton, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Spartanburg, South Carolina
  - Dallas, Texas
  - Laredo, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Argentina (4):
  - Rosario, Santa Fe Province
  - Santa Fé, Santa Fe Province
  - Capital Federal-Buenos Aires
  - Mendoza
- Australia (6):
  - Garran, Australian Capital Territory
  - Camperdown, New South Wales
  - Liverpool, New South Wales
  - Westmead, New South Wales
  - Heidelberg, Victoria
  - Wodonga, Victoria
- Bruxelles - Brussel, Belgium
- Brazil (2):
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
- Canada (5):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Santiago, Chile
- France (10):
  - Bordeaux
  - Caen
  - Lille
  - Lyon
  - Marseille
  - Nantes
  - Paris
  - Strasbourg
  - Toulouse
  - Villejuif
- Germany (10):
  - Mannheim, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Dresden, Saxony
  - Berlin, State of Berlin
- Hungary (3):
  - Budapest
  - Debrecen
  - Zalaegerszeg
- Israel (2):
  - Haifa
  - Tel Aviv
- Italy (6):
  - Milan
  - Modena
  - Pavia
  - Perugia
  - Reggio Emilia
  - Roma
- Nijmegen, Netherlands
- Poland (8):
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Szczecin
  - Warsaw
  - Wroclaw
- Russia (6):
  - Barnaul
  - Kazan'
  - Kirov
  - Moscow
  - Obninsk
  - Saint Petersburg
- South Africa (4):
  - Bloemfontein, Freestate
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (4):
  - Barcelona, Barcelona
  - Cruces/Barakaldo, Bilbao
  - Madrid, Madrid
  - Valencia, Valencia
- Ukraine (5):
  - Donetsk
  - Kharkiv
  - Kiev
  - Lviv
  - Poltava
- United Kingdom (7):
  - Manchester, Manchester
  - Northwood, Middlesex
  - Cardiff, South Glamorgan
  - Glasgow, Stratchclyde
  - Sutton, Surrey
  - Newcastle upon Tyne, Tyne and Wear
  - Birmingham, West Midlands

REFERENCES:
- [Result] Antoun S, Birdsell L, Sawyer MB, Venner P, Escudier B, Baracos VE. Association of skeletal muscle wasting with treatment with sorafenib in patients with advanced renal cell carcinoma: results from a placebo-controlled study. J Clin Oncol. 2010 Feb 20;28(6):1054-60. doi: 10.1200/JCO.2009.24.9730. Epub 2010 Jan 19. PMID 20085939
- [Result] Bellmunt J, Eisen T, Fishman M, Quinn D. Experience with sorafenib and adverse event management. Crit Rev Oncol Hematol. 2011 Apr;78(1):24-32. doi: 10.1016/j.critrevonc.2010.03.006. Epub 2010 Apr 18. PMID 20399677
- [Result] Massard C, Zonierek J, Gross-Goupil M, Fizazi K, Szczylik C, Escudier B. Incidence of brain metastases in renal cell carcinoma treated with sorafenib. Ann Oncol. 2010 May;21(5):1027-31. doi: 10.1093/annonc/mdp411. Epub 2009 Oct 22. PMID 19850637
- [Result] Negrier S, Jager E, Porta C, McDermott D, Moore M, Bellmunt J, Anderson S, Cihon F, Lewis J, Escudier B, Bukowski R. Efficacy and safety of sorafenib in patients with advanced renal cell carcinoma with and without prior cytokine therapy, a subanalysis of TARGET. Med Oncol. 2010 Sep;27(3):899-906. doi: 10.1007/s12032-009-9303-z. Epub 2009 Sep 12. PMID 19757215
- [Result] Pena C, Lathia C, Shan M, Escudier B, Bukowski RM. Biomarkers predicting outcome in patients with advanced renal cell carcinoma: Results from sorafenib phase III Treatment Approaches in Renal Cancer Global Evaluation Trial. Clin Cancer Res. 2010 Oct 1;16(19):4853-63. doi: 10.1158/1078-0432.CCR-09-3343. Epub 2010 Jul 22. PMID 20651059
- [Result] Escudier B, Eisen T, Stadler WM, Szczylik C, Oudard S, Staehler M, Negrier S, Chevreau C, Desai AA, Rolland F, Demkow T, Hutson TE, Gore M, Anderson S, Hofilena G, Shan M, Pena C, Lathia C, Bukowski RM. Sorafenib for treatment of renal cell carcinoma: Final efficacy and safety results of the phase III treatment approaches in renal cancer global evaluation trial. J Clin Oncol. 2009 Jul 10;27(20):3312-8. doi: 10.1200/JCO.2008.19.5511. Epub 2009 May 18. PMID 19451442
- [Result] Eisen T, Oudard S, Szczylik C, Gravis G, Heinzer H, Middleton R, Cihon F, Anderson S, Shah S, Bukowski R, Escudier B; TARGET Study Group. Sorafenib for older patients with renal cell carcinoma: subset analysis from a randomized trial. J Natl Cancer Inst. 2008 Oct 15;100(20):1454-63. doi: 10.1093/jnci/djn319. Epub 2008 Oct 7. PMID 18840822
- [Result] Bukowski R, Cella D, Gondek K, Escudier B; Sorafenib TARGETs Clinical Trial Group. Effects of sorafenib on symptoms and quality of life: results from a large randomized placebo-controlled study in renal cancer. Am J Clin Oncol. 2007 Jun;30(3):220-7. doi: 10.1097/01.coc.0000258732.80710.05. PMID 17551296
- [Result] Escudier B, Eisen T, Stadler WM, Szczylik C, Oudard S, Siebels M, Negrier S, Chevreau C, Solska E, Desai AA, Rolland F, Demkow T, Hutson TE, Gore M, Freeman S, Schwartz B, Shan M, Simantov R, Bukowski RM; TARGET Study Group. Sorafenib in advanced clear-cell renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):125-34. doi: 10.1056/NEJMoa060655. PMID 17215530
- [Result] Kane RC, Farrell AT, Saber H, Tang S, Williams G, Jee JM, Liang C, Booth B, Chidambaram N, Morse D, Sridhara R, Garvey P, Justice R, Pazdur R. Sorafenib for the treatment of advanced renal cell carcinoma. Clin Cancer Res. 2006 Dec 15;12(24):7271-8. doi: 10.1158/1078-0432.CCR-06-1249. PMID 17189398
- [Result] Lamuraglia M, Escudier B, Chami L, Schwartz B, Leclere J, Roche A, Lassau N. To predict progression-free survival and overall survival in metastatic renal cancer treated with sorafenib: pilot study using dynamic contrast-enhanced Doppler ultrasound. Eur J Cancer. 2006 Oct;42(15):2472-9. doi: 10.1016/j.ejca.2006.04.023. Epub 2006 Sep 11. PMID 16965911
- [Derived] Quintanilha JCF, Geyer S, Etheridge AS, Racioppi A, Hammond K, Crona DJ, Pena CE, Jacobson SB, Marmorino F, Rossini D, Cremolini C, Sanoff HK, Abou-Alfa GK, Innocenti F. KDR genetic predictor of toxicities induced by sorafenib and regorafenib. Pharmacogenomics J. 2022 Dec;22(5-6):251-257. doi: 10.1038/s41397-022-00279-3. Epub 2022 Apr 28. PMID 35484400
- [Derived] Quintanilha JCF, Racioppi A, Wang J, Etheridge AS, Denning S, Pena CE, Skol AD, Crona DJ, Lin D, Innocenti F. PIK3R5 genetic predictors of hypertension induced by VEGF-pathway inhibitors. Pharmacogenomics J. 2022 Feb;22(1):82-88. doi: 10.1038/s41397-021-00261-5. Epub 2021 Nov 13. PMID 34775477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From randomization start on 01 Dec 2003 to 31 May 2005 [last subject randomized]. One subject randomized in Placebo did not receive treatment. This study was conducted at 120 centers from 19 countries.
Pre-assignment Details: Enrollment included outpatients with documented unresectable and/or metastatic RCC (Renal Cell Carcinoma), and subjects who had 1 prior systemic therapy for advanced disease on which the subject progressed, at least 1 unidimensional measurable lesion, intermediate or low Motzer risk score, life expectancy of 12 weeks.
Groups:
- Sorafenib (Nexavar, BAY43-9006): Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily).
- Placebo: Subjects received matching placebo tablets administered orally twice a day. [until ~31 May 2005]
- Placebo Randomized, Switch to Sorafenib; Sorafenib Period Only: Subjects received matching placebo tablets administered orally twice a day(as of ~31 May 2005) when after unblinding subjects switched over to receive Sorafenib orally administered as 2 x 200 mg tablets bid (twice daily).
Period: Double-Blind (DB, as of ~31May2005)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Placebo Randomized, Switch to Sorafenib; Sorafenib Period Only
Started | 451 | 452 | 0
Participants Received Treatment | 451 | 451 | 0
Completed | 254 | 299 | 0
Not Completed | 197 | 153 | 0
Not completed — Adverse Event | 22 | 17 | 0
Not completed — Lost to Follow-up | 1 | 6 | 0
Not completed — Withdrawal by Subject | 6 | 11 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Non-compliant with Study medication | 1 | 2 | 0
Not completed — Unknown reason. | 1 | 0 | 0
Not completed — Protocol driven decision point | 0 | 1 | 0
Not completed — entered Open Label (OL); Sorafenib only | 165 | 114 | 0
Not completed — Subject did not receive treatment | 0 | 1 | 0
Period: Open Label-Sorafenib Only [30Jun2008]
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Placebo Randomized, Switch to Sorafenib; Sorafenib Period Only
Started | 254 | 0 (Placebo treatment ended ~ 31May2005. Those who continued, switched to receive Sorafenib.) | 299
Entered OL With Sorafenib Only Phase | 219 | 0 | 216
Completed | 120 | 0 | 143
Not Completed | 134 | 0 | 156
Not completed — Adverse Event | 17 | 0 | 19
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Withdrawal by Subject | 19 | 0 | 9
Not completed — Study terminated by Sponsor | 37 | 0 | 28
Not completed — Per Investigator, not protocol driven | 1 | 0 | 1
Not completed — Switched to commercial drug | 1 | 0 | 1
Not completed — Switched to commercial drug (code error) | 0 | 0 | 3
Not completed — Missing | 3 | 0 | 1
Not completed — No record of treatment discontinuation | 19 | 0 | 9
Not completed — Did not enter OL/ Sorafenib only phase | 35 | 0 | 83

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 451 | 452 | 903
Age, Continuous [Median (Full Range); unit: Years] | 58.0 [19.0 to 86.0] | 59.0 [29.0 to 84.0] | 59.0 [19.0 to 86.0]
Age, Customized [Number; unit: Participants]
  <65 years | 304 | 328 | 632
  >= 65 years | 147 | 124 | 271
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 112 | 248
  Male | 315 | 340 | 655
Motzer Category (Low, intermediate or high) [Number; unit: Participants] — The Motzer score risk factors predicting survival in participants with metastatic RCC are as following: • Low ECOG performance status (PS>2) • High lactate dehydrogenase (>1.5 times upper limit of normal) • Low serum hemoglobin (<lower limit of normal) • High corrected serum calcium (>10 mg/dL) • Absence of prior nephrectomy factors.
  Participants
    Low | 234 | 219 | 453
    Intermediate | 217 | 232 | 449
    Missing | 0 | 1 | 1
ECOG Performance Status (PS) [Number; unit: Participants by scale] — ECOG = Eastern cooperative oncology group PS levels are 0 (Fully active, able to carry on all pre-disease performance), 1 (ambulatory and able to carry out work of a light or sedentary), 2 (Ambulatory and capable of all selfcare but unable to carry out any work activities), 3 (Capable of only limited selfcare, confined to bed or chair more than 50% of awake time), 4 (Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair) and 5 (death).
  Participants by scale
    PS 0 | 219 | 211 | 430
    PS 1 | 223 | 235 | 458
    PS 2 | 7 | 4 | 11
    Missing | 2 | 2 | 4
TNM Classification at study entry [Number; unit: Participants] — TNM=Tumor, primary (T); Nodes, regional lymph nodes (N); Metastasis, distant (M). T0/N0/M0=no evidence of aspect. N1=metastasis in single regional lymph node, M1=distant metastasis. T1=tumor 7 cm or less in greatest dimension limited to kidney. T2= tumor >7 cm in greatest dimension limited to kidney. T3=tumor extends into major veins, invades adrenal gland, or peripheric tissues but not beyond Gerota's fascia. T4=tumor invades beyond Gerota's fascia. [Stage I: T1, N0, M0][Stage II=T2, N0, M0][Stage IV=T4, N0, M0; T4, N1, M0; any T, N2, M0; any T, any N, M1][Stage III=remaining combinations]
  Participants
    Stage III | 18 | 14 | 32
    Stage IV | 433 | 438 | 871
Cancer Subtypes [Number; unit: Participants with carcinoma type] — Histopathological characterization of renal cell carcinomas that subjects had included clear cell, papillary or granular carcinomas. Clear cell renal cell carcinoma is a renal cortical tumor typically characterized by malignant epithelial cells with clear cytoplasm and a compact-alveolar (nested) or acinar growth pattern interspersed with intricate, arborizing vasculature.
  Tumors in which eosinophilic cells predominate were classified as "granular cell" carcinoma.
  Papillary renal cell carcinoma is an uncommon subtype that has distinctive gross, histologic, and cytogenetic features.
  Participants with carcinoma type
    Clear Cell | 449 | 447 | 896
    Papillary | 1 | 3 | 4
    Granular | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Final Overall Survival (OS) - Primary Analysis in the ITT (Intent To Treat) Population
Description: Overall survival determined as the time (days) from the date of randomization at start of study to the date of death, due to any cause. Outcome measure was assessed regularly, i.e. every 3 weeks for the first 24 weeks during treatment and every 4 weeks thereafter and approximately every 3 months during post-treatment.
Time Frame: From start of randomization of the first subject (1Dec2003) until the data cut-off (8Sep2006) for the final OS analysis, approximately 33 months later
Population: Evaluations based on ITT population. Subjects alive at time of analysis were censored at last date of follow-up (FU) (last visit or contact or at data cut-off date). In case of incomplete date, day was missing, day 15 was used.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 451 | 452
days | 542 [500 to 598] | 461 [408 to 526]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Sample size based on primary efficacy endpoint of OS. Clinically meaningful improvement defined as 33.3% improvement in median OS (i.e. HR of 0.75, Sorafenib over Placebo). With overall two-sided alpha of 0.04, 90% power and randomization of 1:1, two formal interim analyses and one final analysis were planned using O'Brien-Fleming type error spending function, and a total of approximately 540 events (deaths) were required for the final analysis; Test type: Superiority or Other; p = 0.146, Log Rank — According to O'Brien-Fleming type alpha spending function and total actual deaths at final analysis, threshold for statistical significance was alpha=0.037 (two-sided); Hazard Ratio (HR) = 0.88, 95% CI [0.74 to 1.04] — Two treatment groups compared using log-rank test (Sorafenib over Placebo) stratified by country and Motzer category

2. Primary Outcome: Final Overall Survival - Secondary Analysis (Placebo Data Censored at 30June2005) in the ITT Population
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Evaluations based on ITT population. Subjects alive at time of analysis were censored at last date of FU (last visit or contact or at data cut-off date). In case of incomplete date, missing day, day 15 was used. Placebo censored at 30June2005, approximate time of crossover of placebo subjects to sorafenib. NA - not estimable due to censored data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 451 | 452
days | 542 [500 to 598] | 436 [385 to NA] — not estimable due to censored data.
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0287, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI [0.62 to 0.97] — Two treatment groups compared using log-rank test (Sorafenib over Placebo) stratified by country and Motzer category

3. Secondary Outcome: Final Progression-Free Survival (PFS) - Independent Radiological Review
Description: PFS determined as the time (days) from the date of randomization at start of study to the actual date of disease progression (PD) (radiological or clinical) or death due to any cause, if death occurred before PD. Outcome measure was assessed approximately every 8 weeks using RECIST v1.0 criteria by independent radiologic review. Radiological PD defined as at least 20% increase in sum of longest diameter (LD) of measured lesions taking as reference smallest sum LD recorded since treatment started or appearance of new lesions.
Time Frame: From start of randomization of the first subject (1Dec2003) until the data cut-off (28Jan2005), approximately 14 months later, tumors assessed every 8 weeks.
Population: Evaluations based on ITT population as of 28Jan2005 data cut; 769 subjects randomized at that time. PFS determined as time from randomization to actual date of disease progression (PD) (radiological or clinical) or death, if death occurred before PD. Subjects without PD or death at time of analysis were censored at last date of tumor assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 384 | 385
days | 167 [139 to 174] | 84 [78 to 91]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; The planned final PFS analysis was to be performed when approximately 363 progressions or deaths (if death occurred before progression) were observed. The analysis had power of 90% to detect a 50% increase in PFS using a two-sided alpha of 0.01; Test type: Superiority or Other; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI [0.35 to 0.55] — Two treatment groups compared using log-rank test (Sorafenib over Placebo) stratified by country and Motzer category

4. Secondary Outcome: Best Overall Response - Independent Radiological Review
Description: Best overall response was determined according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 by independent radiologic review. Categories: complete response (CR, tumor disappears), partial response (PR, sum of lesion sizes decreased), stable disease (SD, steady state of disease), progressive disease (PD, sum of lesion sizes increased) and not evaluated.
Time Frame: as for outcome 3
Population: Evaluations of best overall response based on the valid for response population, where as per protocol, subjects were to have first post-baseline tumor evaluation performed at the end of Cycle 1 (6 weeks post-randomization). Of the ITT population that met this criteria as of the 28Jan2005 data cut, 672 subjects were valid for response.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 335 | 337
percentage of participants
  Complete Response | 0.0 | 0.0
  Partial Response | 2.1 | 0.0
  Stable Disease | 77.9 | 55.2
  Progressive Disease | 8.7 | 30.3
  Not Evaluated | 11.3 | 14.5
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Adjustments for country and Motzer category; Difference in response rates (CR+PR) = -2.1, 95% CI [-3.7 to -0.6] — difference in response rates (CR+PR) = Placebo - Sorafenib

5. Secondary Outcome: Health-related Quality of Life (HRQOL) by FKSI-10 (Functional Assessment of General Therapy Kidney Symptom Index 10) Assessment
Description: Primary Analysis for FKSI-10 patient-reported outcome (PRO) measure defined as longitudinal analysis of mean score over the first 5 treatment cycles. FKSI-10 patient responses for each question range from "0=not at all" to "4=very much" and after reverse coding the range of values for FKSI-10 total score is from 0 to 40; higher score represents better HRQOL.
Time Frame: From start of randomization of the first subject (1Dec2003) until the data cut-off (31May2005), approximately 18 months later, PRO data collected at Day 1 of each cycle and end of treatment.
Population: Evaluations based on ITT population with a PRO assessment. Day 1, Cycle 1 served as baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 451 | 452
Scores on a scale
  Cycle 2, Day 1 | 27.77 (0.23) | 27.78 (0.22)
  Cycle 3, Day 1 | 27.27 (0.22) | 27.28 (0.23)
  Cycle 4, Day 1 | 26.77 (0.25) | 26.78 (0.26)
  Cycle 5, Day 1 | 26.27 (0.30) | 26.28 (0.31)
  Cycles 1-5 (Overall) | 27.19 (0.23) | 27.20 (0.23)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Approximately 200 subjects per group, assuming a 10% drop out rate, were required to detect a 2 point difference between sorafenib and placebo at approximately 80% power with a two-sided alpha of 0.05; Test type: Superiority or Other; p = 0.98, random coefficient model; Random coefficient model adjusted for baseline Motzer score, baseline FKSI-10 score and relative day of FKSI-10 completion

6. Secondary Outcome: Health-related Quality of Life (HRQOL) by Physical Well-Being (PWB) Score of the FACT-G (Functional Assessment of Cancer Therapy-General Version) Assessment
Description: Primary Analysis for FACT-G (using PWB score) patient-reported outcome (PRO) measure defined as longitudinal analysis of mean score over the first 5 treatment cycles. FACT-G (PWB score) patient responses for each question range from "0=not at all" to "4=very much" and after reverse coding the total FACT-G (PWB score) range of values is from 0 to 28; higher score represents better HRQOL.
Time Frame: as for outcome 5
Population: Evaluations based on ITT population with a PRO assessment. Day 1, Cycle 1 served as baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 451 | 452
Scores on a scale
  Cycle 2, Day 1 | 21.21 (0.17) | 21.16 (0.19)
  Cycle 3, Day 1 | 20.77 (0.17) | 20.72 (0.19)
  Cycle 4, Day 1 | 20.33 (0.19) | 20.28 (0.22)
  Cycle 5, Day 1 | 19.89 (0.24) | 19.84 (0.26)
  Cycles 1-5 (Overall) | 20.70 (0.17) | 20.65 (0.19)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.83, random coefficient model; Random coefficient model adjusted for baseline Motzer score, baseline PWB score and relative day of PWB completion

ADVERSE EVENTS:
Time Frame: In addition, 1 participant who was not randomized to double-blind treatment received sorafenib treatment on a compassionate-use basis in the crossover phase and was included in the safety population only.
Description: DIC (disseminated intravascular coagulation), AT (Atrial tachycardia), NOS (not otherwise specified), GI (gastro-intestinal), CTCAE (Common Terminology Criteria for Adverse Events), ANC (absolute neutrophil count), CNS (central nervous system), CN (cranial nerve), GU (genitourinary)
Groups:
- Sorafenib (Nexavar, BAY43-9006)-31May2005 DB: Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily). Double Blind period-31May2005
- Placebo-31May2005 DB: Subjects received matching placebo tablets administered orally twice a day. [until ~31 May 2005]
- Sorafenib (Nexavar, BAY43-9006)-30Jun2008: Sorafenib was to be orally administered as 2 x 200 mg tablets bid (twice daily). Double Blind-30Jun2008. In addition, 1 participant who was not randomized to double-blind treatment received sorafenib treatment on a compassionate-use basis in the open-label/Sorafenib only phase and was included in the safety population only. Participants affected may deviate from double-blind phase due to data update and cleaning.
- Placebo ~31May2005, Then Switched to Sorafenib Only-30Jun2008: Sorafenib period only-30Jun2008: Subjects received matching placebo tablets administered orally twice a day(as of ~31 May 2005) when after unblinding subjects switched over to receive Sorafenib orally administered as 2 x 200 mg tablets bid (twice daily). Open Label/Sorafenib only period-30Jun2008
Arm/Group | Sorafenib (Nexavar, BAY43-9006)-31May2005 DB | Placebo-31May2005 DB | Sorafenib (Nexavar, BAY43-9006)-30Jun2008 | Placebo ~31May2005, Then Switched to Sorafenib Only-30Jun2008
Serious Adverse Events (participants affected / at risk) | 154/451 | 110/451 | 245/452 | 124/216
Other Adverse Events (participants affected / at risk) | 407/451 | 346/451 | 425/452 | 200/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006)-31May2005 DB (N=451) | Placebo-31May2005 DB (N=451) | Sorafenib (Nexavar, BAY43-9006)-30Jun2008 (N=452) | Placebo ~31May2005, Then Switched to Sorafenib Only-30Jun2008 (N=216)
Hemoglobin (Blood and lymphatic system disorders) | 8 | 11 | 16 | 9
Blood - Other (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Platelets (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
DIC (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Edema: Limb (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphatics - Other (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Supraventricular Arrhythmia, Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 3 | 1
Supraventricular Arrhythmia,supraventricular Arrhythmia NOS (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 | 0 | 1 | 1
Supraventricular Arrhythmia, ATrial Tach/Paroxysmal AT (Cardiac disorders) | 1 | 0 | 1 | 1
Supraventricular Arrhythmia, Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 5 | 1 | 0 | 0
Restrictive Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Left Ventricular Diastolic Dysfunction (Cardiac disorders) | 2 | 0 | 2 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertension (Cardiac disorders) | 5 | 0 | 6 | 3
Cardiac Ischemia/Infarction (Cardiac disorders) | 11 | 2 | 18 | 3
Hypotension (Cardiac disorders) | 1 | 0 | 2 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac General - Other (Cardiac disorders) | 2 | 0 | 13 | 9
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 | 0 | 4 | 4
Eyelid Dysfunction (Eye disorders) | 0 | 0 | 1 | 0
Ocular - Other (Eye disorders) | 0 | 1 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 1 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 5 | 2
Dehydration (Gastrointestinal disorders) | 4 | 1 | 6 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 5 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fistula, GI, Colon/Cecum/Appendix (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fistula, GI, Duodenum (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucositis (Functional/Symptomatic), Esophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mucositis (Functional/Symptomatic), Oral Cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Obstruction, GI, Colon (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Obstruction, GI, Duodenum (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Obstruction, GI, Gallbladder (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Obstruction, GI, Ileum (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Obstruction, GI, Small Bowel NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 1
GI - Other (Gastrointestinal disorders) | 3 | 1 | 8 | 4
Perforation, GI, Colon (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Perforation, GI, Small Bowel NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Perforation, GI, Stomach (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stricture, GI, Biliary Tree (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Stricture, GI, Small Bowel NOS (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Ulcer, GI, Duodenum (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 5 | 4 | 2
Death Not Associated With CTCAE Term, Death NOS (General disorders) | 0 | 1 | 3 | 0
Death Not Associated With CTCAE Term, Disease Progression NOS (General disorders) | 11 | 10 | 39 | 32
Death Not Associated With CTCAE Term, Multi-Organ Failure (General disorders) | 0 | 0 | 1 | 1
Death Not Associated With CTCAE Term, Sudden Death (General disorders) | 0 | 1 | 0 | 0
Fever (General disorders) | 4 | 2 | 4 | 2
Fatigue (General disorders) | 7 | 4 | 13 | 6
Weight Loss (General disorders) | 0 | 0 | 1 | 0
Constitutional Symptoms - Other (General disorders) | 10 | 7 | 11 | 6
Pain, Back (General disorders) | 1 | 2 | 5 | 3
Pain, Chest/Thorax NOS (General disorders) | 0 | 1 | 1 | 2
Pain, Chest Wall (General disorders) | 1 | 0 | 1 | 0
Pain, Extremity-Limb (General disorders) | 0 | 5 | 1 | 1
Pain, Tumor Pain (General disorders) | 7 | 4 | 7 | 2
Pain, Abdomen NOS (General disorders) | 4 | 1 | 7 | 4
Pain, Head/Headache (General disorders) | 1 | 2 | 2 | 0
Pain, Joint (General disorders) | 0 | 0 | 1 | 0
Pain, Bone (General disorders) | 3 | 3 | 6 | 4
Pain, Other (General disorders) | 4 | 1 | 3 | 3
Pain, Pelvis (General disorders) | 0 | 0 | 0 | 1
Pain, Neck (General disorders) | 0 | 1 | 0 | 0
Pain, Neuralgia/Peripheral Nerve (General disorders) | 0 | 1 | 0 | 2
Pain, Pain NOS (General disorders) | 1 | 0 | 2 | 0
Flu-Like Syndrome (General disorders) | 0 | 0 | 0 | 1
Tumor Lysis Syndrome (General disorders) | 0 | 0 | 0 | 1
Syndromes - Other (General disorders) | 1 | 0 | 1 | 0
Not Coded Yet (General disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 1 | 2
Liver Dysfunction (Hepatobiliary disorders) | 2 | 2 | 3 | 1
Hepatobiliary - Other (Hepatobiliary disorders) | 1 | 0 | 3 | 3
Pancreatitis (Hepatobiliary disorders) | 2 | 1 | 2 | 2
Allergic Reaction (Immune system disorders) | 0 | 0 | 1 | 0
Allergy - Other (Immune system disorders) | 0 | 0 | 0 | 1
Infection (Documented Clinically), Blood (Infections and infestations) | 1 | 0 | 1 | 1
Infection (Documented Clinically), Bronchus (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Documented Clinically), Catheter-Related (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Documented Clinically), Colon (Infections and infestations) | 1 | 0 | 1 | 0
Infection (Documented Clinically), Lung (Pneumonia) (Infections and infestations) | 2 | 0 | 3 | 0
Infection (Documented Clinically), Meninges (Meningitis) (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Documented Clinically), Skin (Cellulitis) (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Documented Clinically), Urinary Tract NOS (Infections and infestations) | 1 | 0 | 2 | 1
Infection (Documented Clinically), Vein (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Documented Clinically), Wound (Infections and infestations) | 0 | 1 | 1 | 0
Infection With Normal ANC, Appendix (Infections and infestations) | 0 | 0 | 1 | 0
Infection With Normal ANC, Bronchus (Infections and infestations) | 0 | 0 | 0 | 3
Infection With Normal ANC, Catheter-Related (Infections and infestations) | 1 | 0 | 1 | 0
Infection With Normal ANC, Lung (Pneumonia) (Infections and infestations) | 0 | 1 | 0 | 1
Infection With Normal ANC, PANCreas (Infections and infestations) | 0 | 0 | 1 | 0
Infection With Normal ANC, Pelvis NOS (Infections and infestations) | 0 | 0 | 1 | 0
Infection With Normal ANC, Urinary Tract NOS (Infections and infestations) | 0 | 1 | 0 | 0
Opportunistic Infection (Infections and infestations) | 1 | 1 | 0 | 0
Infection - Other (Infections and infestations) | 1 | 1 | 2 | 3
Infection With Unknown ANC, Abdomen NOS (Infections and infestations) | 0 | 0 | 0 | 1
Infection With Unknown ANC, Bronchus (Infections and infestations) | 0 | 0 | 0 | 1
Infection With Unknown ANC, Lung (Pneumonia) (Infections and infestations) | 1 | 1 | 2 | 1
Infection With Unknown ANC, Meninges (Meningitis) (Infections and infestations) | 1 | 0 | 1 | 0
Infection With Unknown ANC, Upper Airway NOS (Infections and infestations) | 0 | 0 | 0 | 1
Infection With Unknown ANC, Urinary Tract NOS (Infections and infestations) | 1 | 0 | 1 | 0
Intraop Injury, Liver (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intraop Injury, Extremity - Upper (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intraop Injury, Bone (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Intraop Injury, Soft Tissue NOS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intraop Injury - Other (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Creatinine (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 6 | 3 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Lipase (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 1
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0
Proteinuria (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 7 | 5 | 12 | 3
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2 | 4 | 7 | 5
Gait/Walking (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle Weakness, Extremity-Lower (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Secondary Malignancy (Possibly Related To Cancer Treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 3 | 1
CNS Ischemia (Nervous system disorders) | 1 | 3 | 7 | 1
Pyramidal Tract Disfunction (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy: Cranial, CN VII Motor-Face; Sensory-Taste (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive DisturbANCe (Nervous system disorders) | 1 | 0 | 1 | 0
Confusion (Nervous system disorders) | 1 | 1 | 3 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2
Speech Impairment (Nervous system disorders) | 0 | 1 | 0 | 1
Involuntary Movement (Nervous system disorders) | 0 | 1 | 0 | 0
Mood Alteration, Depression (Nervous system disorders) | 2 | 0 | 3 | 0
Neuropathy: Motor (Nervous system disorders) | 0 | 0 | 1 | 0
Neurology - Other (Nervous system disorders) | 5 | 7 | 11 | 8
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 2 | 2 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary Electrolyte Wasting (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 8 | 2 | 9 | 4
Renal - Other (Renal and urinary disorders) | 4 | 2 | 13 | 6
Obstruction, GU, Ureter (Renal and urinary disorders) | 0 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 11 | 2
Edema: Larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Airway Obstruction, Bronchus (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 9 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 7 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 21 | 10
Dermatitis, Chemoradiation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Decubitus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dermatology - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Dermatitis, Radiation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
CNS Hemorrhage (Vascular disorders) | 1 | 1 | 2 | 0
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 0 | 0 | 1 | 0
Hemorrhage, GI, Anus (Vascular disorders) | 1 | 0 | 1 | 0
Hemorrhage, GI, Colon (Vascular disorders) | 0 | 0 | 1 | 0
Hemorrhage, GI, Duodenum (Vascular disorders) | 1 | 0 | 2 | 0
Hemorrhage, GI, Stomach (Vascular disorders) | 0 | 0 | 3 | 0
Hemorrhage, GI, Jejunum (Vascular disorders) | 0 | 0 | 1 | 0
Hemorrhage, GI, Lower GI NOS (Vascular disorders) | 0 | 0 | 2 | 0
Hemorrhage, GI, Rectum (Vascular disorders) | 2 | 0 | 2 | 1
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 0 | 2 | 4 | 0
Hemorrhage With Surgery (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage - Other (Vascular disorders) | 3 | 1 | 4 | 2
Hemorrhage Pulmonary, Bronchopulmonary NOS (Vascular disorders) | 3 | 2 | 4 | 2
Hemorrhage Pulmonary, Bronchus (Vascular disorders) | 0 | 2 | 0 | 0
Hemorrhage Pulmonary, Larynx (Vascular disorders) | 0 | 0 | 1 | 0
Hemorrhage Pulmonary, Lung (Vascular disorders) | 1 | 1 | 1 | 0
Hemorrhage Pulmonary, Nose (Vascular disorders) | 1 | 0 | 1 | 2
Hemorrhage Pulmonary, Pleura (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage Pulmonary, Respiratory Tract NOS (Vascular disorders) | 2 | 0 | 3 | 1
Hemorrhage, GU, Uterus (Vascular disorders) | 1 | 0 | 1 | 0
Hemorrhage, GU, Urinary NOS (Vascular disorders) | 1 | 0 | 1 | 1
Thrombosis/Embolism (Vascular Access) (Vascular disorders) | 2 | 0 | 1 | 2
Vascular - Other (Vascular disorders) | 0 | 0 | 4 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 | 5 | 9 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006)-31May2005 DB (N=451) | Placebo-31May2005 DB (N=451) | Sorafenib (Nexavar, BAY43-9006)-30Jun2008 (N=452) | Placebo ~31May2005, Then Switched to Sorafenib Only-30Jun2008 (N=216)
Hemoglobin (Blood and lymphatic system disorders) | 30 | 29 | 61 | 23
Edema: Limb (Blood and lymphatic system disorders) | 28 | 22 | 42 | 16
Hypertension (Cardiac disorders) | 74 | 8 | 101 | 39
Anorexia (Gastrointestinal disorders) | 73 | 57 | 111 | 58
Constipation (Gastrointestinal disorders) | 66 | 48 | 79 | 31
Diarrhea (Gastrointestinal disorders) | 195 | 58 | 244 | 118
Heartburn (Gastrointestinal disorders) | 21 | 10 | 27 | 8
Mucositis (Functional/Symptomatic), Oral Cavity (Gastrointestinal disorders) | 17 | 11 | 27 | 26
Mucositis (Clinical Exam), Oral Cavity (Gastrointestinal disorders) | 30 | 3 | 36 | 11
Nausea (Gastrointestinal disorders) | 102 | 86 | 121 | 42
GI - Other (Gastrointestinal disorders) | 25 | 18 | 37 | 7
Vomiting (Gastrointestinal disorders) | 72 | 51 | 89 | 28
Fever (General disorders) | 36 | 34 | 48 | 16
Insomnia (General disorders) | 16 | 20 | 35 | 9
Fatigue (General disorders) | 162 | 122 | 221 | 86
Weight Loss (General disorders) | 46 | 25 | 102 | 60
Constitutional Symptoms - Other (General disorders) | 38 | 20 | 41 | 19
Sweating (General disorders) | 28 | 17 | 33 | 11
Pain, Back (General disorders) | 33 | 39 | 52 | 17
Pain, Chest/Thorax NOS (General disorders) | 18 | 12 | 26 | 6
Pain, Extremity-Limb (General disorders) | 26 | 20 | 44 | 16
Pain, Tumor Pain (General disorders) | 27 | 20 | 32 | 8
Pain, Abdomen NOS (General disorders) | 46 | 41 | 69 | 23
Pain, Head/Headache (General disorders) | 46 | 26 | 57 | 17
Pain, Joint (General disorders) | 45 | 29 | 59 | 12
Pain, Muscle (General disorders) | 41 | 21 | 48 | 6
Pain, Bone (General disorders) | 33 | 34 | 61 | 23
Pain, Other (General disorders) | 31 | 16 | 60 | 28
Infection - Other (Infections and infestations) | 35 | 26 | 56 | 21
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 23 | 21 | 36 | 12
Dizziness (Nervous system disorders) | 17 | 23 | 24 | 6
Mood Alteration, Depression (Nervous system disorders) | 12 | 16 | 25 | 8
Neuropathy: Sensory (Nervous system disorders) | 59 | 29 | 67 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 64 | 92 | 27
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 25 | 15 | 38 | 11
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 58 | 49 | 94 | 29
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 19 | 1 | 23 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 122 | 15 | 143 | 76
Dry Skin (Skin and subcutaneous tissue disorders) | 50 | 18 | 63 | 22
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 133 | 30 | 156 | 84
Dermatology - Other (Skin and subcutaneous tissue disorders) | 67 | 20 | 84 | 30
Pruritus (Skin and subcutaneous tissue disorders) | 85 | 29 | 90 | 27
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 179 | 70 | 196 | 70
Flushing (Skin and subcutaneous tissue disorders) | 33 | 13 | 40 | 9
Hematoma (Vascular disorders) | 18 | 5 | 23 | 2

LIMITATIONS AND CAVEATS:
Per final PFS data (N=769) study unblinded; placebo-randomized subjects switched to sorafenib ~31May2005 (N=216) that diluted final OS, sorafenib treatment effect. Final ITT, N=903, reported safety data include additional data and cleaning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest.

* Bayer will have up to 30/45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable).
* No publication of single center data should be done prior of publication if multi -center data.